CLINICAL TRIAL: NCT02723773
Title: Efficacy, Safety and Immunogenicity of GSK Biologicals' HZ/su Vaccine GSK1437173A in a Phase IIIb, Open-label, Long-term Follow-up Study (ZOE-LTFU) of Studies 110390/113077 (ZOSTER-006/022) and Assessment of Additional Doses in Older Adults
Brief Title: A Long-term Follow-up Study (ZOE-LTFU) of Two Studies 110390 (ZOSTER-006) and 113077 (ZOSTER-022) to Assess the Efficacy, Safety, and Immunogenicity Persistence of GSK Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine and Assessment of 1 or 2 Additional Doses in Two Subgroups of Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 201190; 2015-001778-17 (EudraCT Number)
Record Dates: First submitted 2016-03-10; First posted 2016-03-30 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Herpes Zoster; Herpes Zoster Vaccine
Keywords: Efficacy; Immunogenicity; Safety; Adults; Herpes zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LTFU Group (No Intervention): Participants who received at least 1 dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study were followed up for long-term vaccine efficacy and safety.
- 1-Additional Dose Group (Experimental): Participants who received 2 doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies received 1 additional dose of the HZ/su vaccine at Month 0 in the current ZOSTER-049:EXT 006-022 study.
  Interventions: Biological: Herpes Zoster Vaccine GSK1437173A
- Revaccination Group (Experimental): Participants who received 2 doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies were revaccinated with 2 additional doses of the HZ/su vaccine at Month 0 and Month 2 in the current ZOSTER-049:EXT 006-022 study.
  Interventions: Biological: Herpes Zoster Vaccine GSK1437173A
- Control Group (No Intervention): Participants who received 2 doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study, but who served as a control for the 2 groups that received 1 or 2 additional doses (1-Additional Dose Group and Revaccination Group).

INTERVENTIONS:
Biological: Herpes Zoster Vaccine GSK1437173A — Intramuscular injection
  Arms: 1-Additional Dose Group; Revaccination Group

SUMMARY:
The purpose of this study was a long-term follow-up of the two studies 110390 and 113077 (ZOSTER-006/022) to assess the efficacy, safety, and immunogenicity persistence of GSK Biologicals' Herpes Zoster subunit (HZ/su) vaccine and included an assessment of 1 or 2 additional doses in two subgroups of older adults.

DETAILED DESCRIPTION:
This is the long-term follow-up study (ZOE-LTFU) of studies 110390 and 113077 (ZOSTER-006/022) to assess the prophylactic efficacy, safety, and immunogenicity persistence of GSK Biologicals' Herpes Zoster subunit (HZ/su) vaccine and included an assessment of 1 or 2 additional doses on a 0 or 0, 2-month schedule in two subgroups of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits, ability to have scheduled contacts to allow evaluation during the study). Or subjects with a caregiver who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, availability for follow-up contacts).
* Written informed consent obtained from the subject prior to performance of any study specific procedure.
* Subject who participated in ZOSTER-006 or ZOSTER-022 studies and received at least one dose of HZ/su vaccine.

Additional inclusion criteria for the 1-Additional Dose Revaccination and Control groups, ONLY:

* Female subjects of non-childbearing potential may be enrolled in this study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in this study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (pharmaceutical product or device) at the time of enrolment or planned use during the study period.
* Previous vaccination against Varicella Zoster Virus (VZV) or HZ and/or planned administration during the study of a VZV or HZ vaccine (including an investigational or non-registered vaccine other than the HZ/su vaccine administered in studies ZOSTER-006/022).
* Chronic administration (defined as ≥ 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting six months prior to Visit Month 0 of study ZOSTER-049 or expected administration at any time during the study period. For corticosteroids, this will mean prednisone ≥ 20 mg/day or equivalent. A prednisone dose of < 20 mg/day is allowed. Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration of long-acting immune-modifying drugs (e.g., infliximab, rituximab) within 6 months prior to Visit Month 0 of study ZOSTER-049 or expected administration at any time during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, human immunodeficiency virus [HIV] infection) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders).
* Administration of immunoglobulins and/or any blood products within 3 months prior to Visit Month 0 of study ZOSTER-049 or planned administration during the study period.
* Prolonged use (> 14 consecutive days) of oral and/or parenteral antiviral agents that are active against VZV (acyclovir, valacyclovir, famciclovir, etc. ) and planned to be used during the study period for an indication other than to treat suspected or confirmed HZ or an HZ-related complication (topical use of these antiviral agents is allowed).
* Important underlying illness that in the opinion of the investigator would be expected to interfere significantly during the study.

Additional exclusion criteria for the 1-Additional Dose Revaccination and Control groups, only:

* Subjects who experienced an SAE from first vaccination in the previous ZOSTER-006/022 studies to enrolment in study ZOSTER-049 that was considered related to study vaccine by either the investigator or the sponsor.
* Subjects with a new onset of a pIMD or exacerbation of a pIMD from first vaccination in the previous ZOSTER-006/022 studies to enrolment in study ZOSTER-049.
* Use of any investigational or non-registered product (pharmaceutical product or device) within 30 days preceding the first dose of study vaccine or planned use during the study period.
* Administration or planned administration of any other immunizations within 30 days before the first study vaccination or scheduled within 30 days after study vaccination. However, licensed non-replicating vaccines (i.e., inactivated and subunit vaccines, including inactivated and subunit influenza vaccines for seasonal or pandemic flu, with or without adjuvant) may be administered up to 8 days prior to each dose and/or at least 14 days after any dose of study vaccine.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine. Additionally, consider allergic reactions to other material or equipment related to study participation (such as materials that may possibly contain latex-gloves, syringes, etc.). Please note, the vaccine and vials in this study do not contain latex.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions (if of childbearing potential).
* Previous episode/history of HZ.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7539 (Actual)
Dates: Start 2016-04-16 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (133):
- United States (21):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Wadsworth, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Newport News, Virginia
- Australia (3):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Geelong, Victoria
- Brazil (4):
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Curitiba
  - GSK Investigational Site, CuritibaPR
  - GSK Investigational Site, São Paulo
- Canada (11):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Hradec Králové
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (11):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Château-Gontier
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Montrevault
  - GSK Investigational Site, Muret
  - GSK Investigational Site, Mûrs-Erigné
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Segré
  - GSK Investigational Site, Tours
- Germany (26):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Dachau
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Flörsheim
  - GSK Investigational Site, Freiberg
  - GSK Investigational Site, Goch
  - GSK Investigational Site, Güglingen
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Köthen
  - GSK Investigational Site, Künzing
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Lübeck
  - GSK Investigational Site, Magdeburg
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Mannheim
  - GSK Investigational Site, München
  - GSK Investigational Site, Rednitzhembach
  - GSK Investigational Site, Rhaunen
  - GSK Investigational Site, Tübingen
  - GSK Investigational Site, Wallerfing
  - GSK Investigational Site, Wangen
  - GSK Investigational Site, Weinheim
  - GSK Investigational Site, Witten
  - GSK Investigational Site, Würzburg
- Hong Kong (2):
  - GSK Investigational Site, Kwun Tong Kowloon
  - GSK Investigational Site, Shatin
- Italy (5):
  - GSK Investigational Site, Chieti
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Monza MB
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Sassari
- Japan (3):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Tokyo
- Mexico (2):
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Zapopan Jalisco
- South Korea (5):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Bucheon-si Kyunggi-do 14584
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Alcover Tarragona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Hostalets de Balenya Ba
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Peralada Girona
  - GSK Investigational Site, Valencia
- Sweden (11):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
  - GSK Investigational Site, Vällingby
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tau-Yuan
- United Kingdom (6):
  - GSK Investigational Site, Atherstone Warwickshire
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Bradford on Avon Wiltsh
  - GSK Investigational Site, Broughshane
  - GSK Investigational Site, Chorley
  - GSK Investigational Site, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Strezova A, Diez Domingo J, Cunningham AL, Eto T, Andrews C, Arns C, Choo EJ, Hui DSC, Icardi G, McNeil SA, Poder A, Kosina P, Rombo L, Schwarz TF, Tinoco JC, Yu CJ, Wang J, Soni J, Tsang M, Leon R, Mwakingwe-Omari A; Zoster-049 Study Group. Final analysis of the ZOE-LTFU trial to 11 years post-vaccination: efficacy of the adjuvanted recombinant zoster vaccine against herpes zoster and related complications. EClinicalMedicine. 2025 May 9;83:103241. doi: 10.1016/j.eclinm.2025.103241. eCollection 2025 May. PMID 40630610
- [Derived] Giannelos N, Curran D, Matthews S, Carrico J, Cunningham AL. The Potential Impact of Increased Recombinant Zoster Vaccine Uptake in Older Adults Worldwide. Infect Dis Ther. 2025 Jun;14(6):1327-1341. doi: 10.1007/s40121-025-01161-y. Epub 2025 May 21. PMID 40399558
- [Derived] Boutry C, Hastie A, Diez-Domingo J, Tinoco JC, Yu CJ, Andrews C, Beytout J, Caso C, Cheng HS, Cheong HJ, Choo EJ, Curiac D, Di Paolo E, Dionne M, Eckermann T, Esen M, Ferguson M, Ghesquiere W, Hwang SJ, Avelino-Silva TJ, Kosina P, Liu CS, Markkula J, Moeckesch B, Murta de Oliveira C, Park DW, Pauksens K, Pirrotta P, Plassmann G, Pretswell C, Rombo L, Salaun B, Sanmartin Berglund J, Schenkenberger I, Schwarz T, Shi M, Ukkonen B, Zahaf T, Zerbini C, Schuind A, Cunningham AL; Zoster-049 Study Group. The Adjuvanted Recombinant Zoster Vaccine Confers Long-Term Protection Against Herpes Zoster: Interim Results of an Extension Study of the Pivotal Phase 3 Clinical Trials ZOE-50 and ZOE-70. Clin Infect Dis. 2022 Apr 28;74(8):1459-1467. doi: 10.1093/cid/ciab629. PMID 34283213

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potentially eligible participants who participated and received at least one dose of the HZ/su vaccine in the ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229) primary studies were contacted and considered for entry in the current ZOSTER-049:EXT 006-022 (NCT02723773) study.
Pre-assignment Details: Out of the 7534 participants enrolled in the current ZOSTER-049 EXT:006-022 study, 5 participants originally enrolled in the Long-term follow-up (LTFU) group were eliminated due to data modification post-investigator signature, and hence 7529 participants were included in the Total Vaccinated Cohort and started the study.
Period: Overall Study
Arm/Group | LTFU Group | 1-Additional Dose Group | Revaccination Group | Control Group
Started | 7289 | 61 | 60 | 119
Completed | 5570 | 52 | 51 | 97
Not Completed | 1719 | 9 | 9 | 22
Not completed — Adverse Event | 934 | 3 | 1 | 9
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 360 | 5 | 6 | 10
Not completed — Migrated/moved from study area | 37 | 0 | 0 | 1
Not completed — Lost to Follow-up | 198 | 0 | 0 | 0
Not completed — Other | 189 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LTFU Group | 1-Additional Dose Group | Revaccination Group | Control Group | Total
Number analyzed (Participants) | 7289 | 61 | 60 | 119 | 7529
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.6 (9.4) | 70.4 (9.2) | 70.2 (9.4) | 70.2 (8.6) | 72.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4432 | 30 | 36 | 69 | 4567
  Male | 2857 | 31 | 24 | 50 | 2962
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 66 | 0 | 0 | 0 | 66
  Asian - East Asian Heritage | 1115 | 0 | 0 | 0 | 1115
  Asian - Japanese Heritage | 265 | 0 | 0 | 0 | 265
  Other, Deidentified | 5843 | 61 | 60 | 119 | 6083

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Having at Least One Confirmed Herpes Zoster (HZ) Case During the Total Duration of ZOSTER-049:EXT 006-022 Study, Overall
Description: A suspected case of HZ is defined as a new unilateral rash accompanied by pain and no alternative diagnosis. A confirmed case of HZ was diagnosed by Polymerase Chain Reaction (PCR) and/or by HZ Ascertainment Committee (HZAC) determination, as per the algorithm pre-specified in the protocol.
  As pre-specified in the protocol:
  * due to the high VE observed in ZOSTER-006/022 studies, recipients of placebo in both studies were offered cross-vaccination with HZ/su. Since there was no placebo group in this study, historic controls were used for VE assessment. Incidence rates estimations on Historical Control group were done by utilizing Poisson regression model using placebo data from ZOSTER-006/022 studies to obtain the coefficients by age ranges.
  * the participants in Control group were a subset of LTFU group that were randomized to serve as control for those who were vaccinated in this study, otherwise they were treated similarly as LTFU group, hence LTFU and Control groups were combined.
Time Frame: During the total duration of ZOSTER-049:EXT 006-022 study (From Month 0 to Month 72)
Population: The analysis was performed on the Modified Total Vaccinated cohort (mTVC) - LTFU+Control group, which included all participants in the LTFU and Control groups combined, with efficacy data available for the specified analysis during the specified period, minus those participants who were not administered with the second vaccination during the ZOSTER-006/022 studies, or who developed a confirmed case of HZ prior to 1 month after the second vaccination in the ZOSTER-006/022 studies.
Measure: Count of Participants; unit: Participants
Groups:
- LTFU+Control >=50YOA Group: Participants 50 years of age or above (>=50 YOA) (at the time of primary vaccination in the ZOSTER-006/022 studies) who received at least one dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study, i.e., combined group of LTFU group and Control group in the current ZOSTER-049 :EXT 006-022 study.
- Historical Control >=50 YOA Group: Hypothetical control group formed by using incidence rates estimated from actual placebo data in the ZOSTER-006/022 primary studies collected from participants >=50 YOA (at time of primary vaccination in ZOSTER-006/022 studies).
Arm/Group | LTFU+Control >=50YOA Group | Historical Control >=50 YOA Group
Number analyzed (Participants) | 7258 | 7258
Participants | 69 | 341
Statistical Analysis 1: Comparison: LTFU+Control >=50YOA Group vs Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between LTFU+Control >=50 YOA Group and Historical Control >=50 YOA Group; Test type: Other — The statistical analyses performed for the study objectives were descriptive. No success criteria were defined for the statistical analyses conducted in this study; Poisson regression method; Vaccine efficacy = 79.77, 95% CI 2-sided [73.72 to 84.61] — VE=1 - the relative risk (RR). RR=the ratio of the incidence rates of LTFU+Control >=50YOA Group over Historical Control >=50YOA Group. The VE of HZ/su vaccine against HZ in this study was descriptively summarized by age strata and overall

2. Secondary Outcome: Number of Participants Having at Least One Confirmed HZ Case During the Total Duration of ZOSTER-049:EXT 006-022 Study, by Age Ranges
Description: A suspected case of HZ is defined as a new unilateral rash accompanied by pain and no alternative diagnosis. A confirmed case of HZ was diagnosed by PCR and/or by the HZAC determination, as per the algorithm pre-specified in the protocol. The age ranges assessed were: 50-59 YOA, 60-69 YOA, >=60 YOA and >=70 YOA at time of primary vaccination in ZOSTER-006/022 studies.
Time Frame: During the total duration of ZOSTER-049:EXT 006-022 study (From Month 0 to Month 72)
Population: The analysis was performed on the mTVC - LTFU+Control group, which included all participants in the LTFU and Control groups combined, with efficacy data available for the specified analysis and age ranges during the specified period, minus those participants who were not administered with the second vaccination during the ZOSTER-006/022 studies, or who developed a confirmed case of HZ prior to 1 month after the second vaccination in the ZOSTER-006/022 studies.
Measure: Count of Participants; unit: Participants
Groups:
- LTFU+Control 50-59 YOA Group: Participants between 50 and 59 YOA (at time of primary vaccination in ZOSTER-006/022 studies) who received at least one dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study, i.e., combined group of LTFU group and Control group in the current ZOSTER-049:EXT 006-022 study.
- LTFU+Control 60-69 YOA Group: Participants between 60 and 69 YOA (at time of primary vaccination in ZOSTER-006/022 studies) who received at least one dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study, i.e., combined group of LTFU group and Control group in the current ZOSTER-049:EXT 006-022 study.
- LTFU+Control >=60 YOA Group: Participants >=60 YOA (at time of primary vaccination in ZOSTER-006/022 studies) who received at least one dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study, i.e., combined group of LTFU group and Control group in the current ZOSTER-049:EXT 006-022 study.
- LTFU+Control >=70 YOA Group: Participants >=70 YOA (at time of primary vaccination in ZOSTER-006/022 studies) who received at least one dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study, i.e., combined group of LTFU group and Control group in the current ZOSTER-049:EXT 006-022 study.
- Historical Control 50-59 YOA Group: Hypothetical control group formed by using incidence rates estimated from actual placebo data in the ZOSTER-006/022 primary studies collected from participants between 50 and 59 YOA (at time of primary vaccination in ZOSTER-006/022 studies).
- Historical Control 60-69 YOA Group: Hypothetical control group formed by using incidence rates estimated from actual placebo data in the ZOSTER-006/022 primary studies collected from participants between 60 and 69 YOA (at time of primary vaccination in ZOSTER-006/022 studies).
- Historical Control >=60 YOA Group: Hypothetical control group formed by using incidence rates estimated from actual placebo data in the ZOSTER-006/022 primary studies collected from participants >=60 YOA (at time of primary vaccination in ZOSTER-006/022 studies).
- Historical Control >=70 YOA Group: Hypothetical control group formed by using incidence rates estimated from actual placebo data in the ZOSTER-006/022 primary studies collected from participants >=70 YOA (at time of primary vaccination in ZOSTER-006/022 studies).
Arm/Group | LTFU+Control 50-59 YOA Group | LTFU+Control 60-69 YOA Group | LTFU+Control >=60 YOA Group | LTFU+Control >=70 YOA Group | Historical Control 50-59 YOA Group | Historical Control 60-69 YOA Group | Historical Control >=60 YOA Group | Historical Control >=70 YOA Group
Number analyzed (Participants) | 2043 | 1242 | 5215 | 3973 | 2043 | 1242 | 5215 | 3973
Participants | 12 | 9 | 57 | 48 | 90 | 70 | 249 | 179
Statistical Analysis 1: Comparison: LTFU+Control 50-59 YOA Group vs Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between LTFU+Control 50-59 YOA Group and Historical Control 50-59 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 86.67, 95% CI 2-sided [75.55 to 93.36] — VE = 1 - RR. RR = the ratio of the incidence rates of LTFU+Control 50-59 YOA Group over Historical Control 50-59 YOA Group. The VE of HZ/su vaccine against HZ in this study was descriptively summarized by age strata and overall
Statistical Analysis 2: Comparison: LTFU+Control 60-69 YOA Group vs Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between LTFU+Control 60-69 YOA Group and Historical Control 60-69 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 87.14, 95% CI 2-sided [74.17 to 94.35] — VE = 1 - RR. RR = the ratio of the incidence rates of LTFU+Control 60-69 YOA Group over Historical Control 60-69 YOA Group. The VE of HZ/su vaccine against HZ in this study was descriptively summarized by age strata and overall
Statistical Analysis 3: Comparison: LTFU+Control >=60 YOA Group vs Historical Control >=60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between LTFU+Control >=60 YOA Group and Historical Control >=60 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 77.11, 95% CI 2-sided [69.37 to 83.14] — VE = 1 - RR. RR = the ratio of the incidence rates of LTFU+Control >=60 YOA Group over Historical Control >=60 YOA Group. The VE of HZ/su vaccine against HZ in this study was descriptively summarized by age strata and overall
Statistical Analysis 4: Comparison: LTFU+Control >=70 YOA Group vs Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between LTFU+Control >=70 YOA Group and Historical Control >=70 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 73.18, 95% CI 2-sided [62.94 to 80.92] — VE = 1 - RR. RR = the ratio of the incidence rates of LTFU+Control >=70 YOA Group over Historical Control >=70 YOA Group. The VE of HZ/su vaccine against HZ in this study was descriptively summarized by age strata and overall

3. Secondary Outcome: Number of Participants Having at Least One Confirmed HZ Case From One Month Post-Dose 2 in ZOSTER-006/022 Studies Until the End of ZOSTER-049:EXT 006-022 Study, Overall and by Age Ranges
Description: A suspected case of HZ is defined as a new unilateral rash accompanied by pain and no alternative diagnosis. A confirmed case of HZ was diagnosed by PCR and/or by the HZAC determination, as per the algorithm pre-specified in the protocol. The age ranges assessed were: >=50 YOA (overall), 50-59 YOA, 60-69 YOA, >=60 YOA and >=70 YOA at time of primary vaccination in ZOSTER-006/022 studies.
  As pre-specified in the protocol:
  - participants from the Placebo groups in the ZOSTER-006/022 studies for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start and from the hypothetical Historical control group in the ZOSTER-049:EXT 006-022 study for Year 6 and onwards were combined in the Placebo/Historical control group.
Time Frame: From one month post-Dose 2 (Month 3) in ZOSTER-006/022 primary studies until the end of ZOSTER-049:EXT 006-022 study (Month 72), a period of approximately 12 years
Population: The analysis was performed on the mTVC pooled, which included participants from the mTVC in ZOSTER-006/-022 studies and participants from the mTVC in ZOSTER-049:EXT 006-022 study with efficacy data available for the specified analysis and age ranges during the specified period.
Measure: Count of Participants; unit: Participants
Groups:
- HZ/su >=50 YOA Group: Participants >=50 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received 2 doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies, among which participants who did not enroll in the current ZOSTER-049:EXT 006-022 study only contributed to data for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start.
- HZ/su 50-59 YOA Group: Participants between 50 and 59 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received 2 doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies, among which participants who did not enroll in the current ZOSTER-049:EXT 006-022 study only contributed to data for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start.
- HZ/su 60-69 YOA Group: Participants between 60 and 69 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received 2 doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies, among which participants who did not enroll in the current ZOSTER-049:EXT 006-022 study only contributed to data for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start.
- HZ/su >=60 YOA Group: Participants >=60 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received 2 doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies, among which participants who did not enroll in the current ZOSTER-049:EXT 006-022 study only contributed to data for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start.
- HZ/su >=70 YOA Group: Participants >=70 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received 2 doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies, among which participants who did not enroll in the current ZOSTER-049:EXT 006-022 study only contributed to data for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start.
- Placebo/Historical Control >=50 YOA Group: Participants >=50 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) from the Placebo groups in the ZOSTER-006/022 primary studies for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start and from the hypothetical Historical control group in the current ZOSTER-049:EXT 006-022 study for Year 6 and onwards were combined into this group.
- Placebo/Historical Control 50-59 YOA Group: Participants between 50 and 59 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) from the Placebo groups in the ZOSTER-006/022 primary studies for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start and from the hypothetical Historical control group in the current ZOSTER-049:EXT 006-022 study for Year 6 and onwards were combined into this group.
- Placebo/Historical Control 60-69 YOA Group: Participants between 60 and 69 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) from the Placebo groups in the ZOSTER-006/022 primary studies for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start and from the hypothetical Historical control group in the current ZOSTER-049:EXT 006-022 study for Year 6 and onwards were combined into this group.
- Placebo/Historical Control >= 60 YOA Group: Participants >=60 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) from the Placebo groups in the ZOSTER-006/022 primary studies for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start and from the hypothetical Historical control group in the current ZOSTER-049:EXT 006-022 study for Year 6 and onwards were combined into this group.
- Placebo/Historical Control >=70 YOA Group: Participants >=70 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) from the Placebo groups in the ZOSTER-006/022 primary studies for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start and from the hypothetical Historical control group in the current ZOSTER-049:EXT 006-022 study for Year 6 and onwards were combined into this group.
Arm/Group | HZ/su >=50 YOA Group | HZ/su 50-59 YOA Group | HZ/su 60-69 YOA Group | HZ/su >=60 YOA Group | HZ/su >=70 YOA Group | Placebo/Historical Control >=50 YOA Group | Placebo/Historical Control 50-59 YOA Group | Placebo/Historical Control 60-69 YOA Group | Placebo/Historical Control >= 60 YOA Group | Placebo/Historical Control >=70 YOA Group
Number analyzed (Participants) | 13881 | 3491 | 2140 | 10390 | 8250 | 14035 | 3523 | 2166 | 10512 | 8346
Participants | 101 | 16 | 12 | 85 | 73 | 818 | 193 | 160 | 623 | 463
Statistical Analysis 1: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control 50 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 87.73, 95% CI 2-sided [84.89 to 90.12] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su >=50 YOA Group over Placebo/Historical Control >=50 YOA Group. The VE of HZ/su vaccine against HZ in this study was descriptively summarized by age strata and overall
Statistical Analysis 2: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 91.74, 95% CI 2-sided [86.25 to 95.37] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su 50-59 YOA Group over Placebo/Historical Control 50-59 YOA Group. The VE of HZ/su vaccine against HZ in this study was descriptively summarized by age strata and overall
Statistical Analysis 3: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 92.57, 95% CI 2-sided [86.66 to 96.24] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su 60-69 YOA Group over Placebo/Historical Control 60-69 YOA Group. The VE of HZ/su vaccine against HZ in this study was descriptively summarized by age strata and overall
Statistical Analysis 4: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 86.45, 95% CI 2-sided [82.98 to 89.33] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su >=60 YOA Group over Placebo/Historical Control >=60 YOA Group. The VE of HZ/su vaccine against HZ in this study was descriptively summarized by age strata and overall
Statistical Analysis 5: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 84.33, 95% CI 2-sided [79.91 to 87.93] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su >=70 YOA Group over Placebo/Historical Control >=70 YOA Group. The VE of HZ/su vaccine against HZ in this study was descriptively summarized by age strata and overall

4. Secondary Outcome: Number of Participants Having at Least One Confirmed HZ Case Over the Follow-up Years From One Month Post-Dose 2 in ZOSTER-006/022 Studies Until the End of ZOSTER-049:EXT 006-022 Study, Overall and by Age Ranges
Description: A suspected case of HZ is defined as a new unilateral rash accompanied by pain and no alternative diagnosis. A confirmed case of HZ was diagnosed by PCR and/or by the HZAC determination, as per the algorithm pre-specified in the protocol. The age ranges assessed were: >=50 YOA (overall), 50-59 YOA, 60-69 YOA, >=60 YOA and >=70 YOA at time of primary vaccination in ZOSTER-006/022 studies.
  Confirmed HZ cases data was not collected for the participants included in the HZ/su and Placebo/Historical control groups during Year 5, as this was a gap year between end of ZOSTER-006/-022 studies and start of ZOSTER-049:EXT-006-022 study.
  Results from the ZOSTER-006/022 studies were pooled for each year after vaccination with methods used in these studies. For overlapping years between ZOSTER-006/022 studies and this study, all the data were pooled. For the non-overlapping years only the data from ZOSTER-049:EXT 006-022 study was used.
Time Frame: Over the follow-up years (Year 1, Year 2, Year 3, Year 4, Year 6, Year 7, Year 8, Year 9, Year 10 and Year 11) from one month post-Dose 2 (Month 3) in ZOSTER-006/022 primary studies until the end of ZOSTER-049:EXT 006-022 study (Month 72)
Population: The analysis was performed on the mTVC pooled, which included participants from the mTVC in ZOSTER-006/-022 studies and participants from the mTVC in ZOSTER-049:EXT 006-022 study with efficacy data available for the specified analysis and age ranges during the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su >=50 YOA Group | HZ/su 50-59 YOA Group | HZ/su 60-69 YOA Group | HZ/su >=60 YOA Group | HZ/su >=70 YOA Group | Placebo/Historical Control >=50 YOA Group | Placebo/Historical Control 50-59 YOA Group | Placebo/Historical Control 60-69 YOA Group | Placebo/Historical Control >= 60 YOA Group | Placebo/Historical Control >=70 YOA Group
Number analyzed (Participants) | 13881 | 3491 | 2140 | 10390 | 8250 | 14035 | 3523 | 2166 | 10512 | 8346
Participants
  Year 1 | 3 | 1 | 0 | 2 | 2 | 130 | 31 | 16 | 99 | 83
  Year 2: number analyzed (Participants) | 13569 | 3421 | 2109 | 10148 | 8039 | 13564 | 3427 | 2113 | 10137 | 8024
  Year 2 | 10 | 2 | 1 | 8 | 7 | 136 | 27 | 22 | 109 | 87
  Year 3: number analyzed (Participants) | 13185 | 3371 | 2078 | 9814 | 7736 | 13074 | 3351 | 2062 | 9723 | 7661
  Year 3 | 9 | 0 | 0 | 9 | 9 | 116 | 29 | 29 | 87 | 58
  Year 4: number analyzed (Participants) | 12757 | 3301 | 2030 | 9456 | 7426 | 12517 | 3272 | 1978 | 9245 | 7267
  Year 4 | 10 | 1 | 2 | 9 | 7 | 95 | 16 | 23 | 79 | 56
  Year 6: number analyzed (Participants) | 7258 | 2043 | 1242 | 5215 | 3973 | 7258 | 2043 | 1242 | 5215 | 3973
  Year 6 | 10 | 2 | 1 | 8 | 7 | 62 | 16 | 13 | 47 | 35
  Year 7: number analyzed (Participants) | 7083 | 2020 | 1222 | 5063 | 3841 | 7083 | 2020 | 1222 | 5063 | 3841
  Year 7 | 10 | 1 | 2 | 9 | 7 | 61 | 15 | 13 | 46 | 33
  Year 8: number analyzed (Participants) | 6857 | 1998 | 1198 | 4859 | 3661 | 6857 | 1998 | 1198 | 4859 | 3661
  Year 8 | 10 | 2 | 2 | 8 | 6 | 58 | 15 | 13 | 43 | 31
  Year 9: number analyzed (Participants) | 6627 | 1977 | 1181 | 4650 | 3469 | 6627 | 1977 | 1181 | 4650 | 3469
  Year 9 | 15 | 5 | 3 | 10 | 7 | 57 | 15 | 11 | 42 | 29
  Year 10: number analyzed (Participants) | 6239 | 1908 | 1122 | 4331 | 3209 | 6239 | 1908 | 1122 | 4331 | 3209
  Year 10 | 15 | 0 | 1 | 15 | 14 | 53 | 15 | 10 | 38 | 27
  Year 11: number analyzed (Participants) | 5849 | 1883 | 1075 | 3966 | 2891 | 5849 | 1883 | 1075 | 3966 | 2891
  Year 11 | 9 | 2 | 0 | 7 | 7 | 50 | 15 | 10 | 34 | 25
Statistical Analysis 1: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group over Year 1; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 97.68, 95% CI 2-sided [93.07 to 99.53] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group over Year 1; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 96.76, 95% CI 2-sided [80.57 to 99.92] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group over Year 1; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 100.00, 95% CI 2-sided [79.32 to 100.00] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 4: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group over Year 1; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 97.97, 95% CI 2-sided [92.46 to 99.76] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 5: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group over Year 1; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 97.57, 95% CI 2-sided [90.96 to 99.71] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 6: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group over Year 2; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 92.69, 95% CI 2-sided [86.15 to 96.57] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group over Year 2; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 92.66, 95% CI 2-sided [70.78 to 99.15] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 8: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group over Year 2; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 95.49, 95% CI 2-sided [72.11 to 99.89] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 9: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group over Year 2; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 92.71, 95% CI 2-sided [85.13 to 96.93] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 10: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group over Year 2; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 92.01, 95% CI 2-sided [82.82 to 96.88] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 11: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group over Year 3; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 92.36, 95% CI 2-sided [84.98 to 96.59] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group over Year 3; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 100.00, 95% CI 2-sided [89.20 to 100.00] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 13: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group over Year 3; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 100.00, 95% CI 2-sided [89.39 to 100.00] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 14: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group over Year 3; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 89.84, 95% CI 2-sided [79.81 to 95.51] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 15: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group over Year 3; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 84.74, 95% CI 2-sided [68.99 to 93.35] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 16: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group over Year 4; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 89.75, 95% CI 2-sided [80.31 to 95.24] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 17: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group over Year 4; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 93.88, 95% CI 2-sided [60.62 to 99.85] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 18: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group over Year 4; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 91.62, 95% CI 2-sided [66.10 to 99.04] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 19: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group over Year 4; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 88.96, 95% CI 2-sided [77.96 to 95.13] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 20: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group over Year 4; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 87.86, 95% CI 2-sided [73.30 to 95.33] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 21: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group over Year 6; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 83.87, 95% CI 2-sided [68.31 to 92.63] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 22: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group over Year 6; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 87.50, 95% CI 2-sided [46.83 to 98.61] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 23: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group over Year 6; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 92.31, 95% CI 2-sided [48.79 to 99.82] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 24: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group over Year 6; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 82.98, 95% CI 2-sided [63.64 to 93.05] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 25: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group over Year 6; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 80.00, 95% CI 2-sided [54.30 to 92.50] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 26: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group over Year 7; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 83.61, 95% CI 2-sided [67.76 to 92.51] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 27: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group over Year 7; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 93.33, 95% CI 2-sided [56.67 to 99.84] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 28: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group over Year 7; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 84.62, 95% CI 2-sided [32.04 to 98.31] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 29: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group over Year 7; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 80.43, 95% CI 2-sided [59.54 to 91.58] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 30: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group over Year 7; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 78.79, 95% CI 2-sided [51.24 to 92.08] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 31: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group over Year 8; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 82.76, 95% CI 2-sided [65.98 to 92.14] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 32: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group over Year 8; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 86.67, 95% CI 2-sided [42.67 to 98.52] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 33: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group over Year 8; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 84.62, 95% CI 2-sided [32.04 to 98.31] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 34: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group over Year 8; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 81.40, 95% CI 2-sided [59.97 to 92.45] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 35: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group over Year 8; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 80.65, 95% CI 2-sided [52.91 to 93.40] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 36: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group over Year 9; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 73.68, 95% CI 2-sided [52.89 to 86.16] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 37: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group over Year 9; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 66.67, 95% CI 2-sided [3.52 to 90.52] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 38: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group over Year 9; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 72.73, 95% CI 2-sided [-3.24 to 95.11] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 39: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group over Year 9; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 76.19, 95% CI 2-sided [51.78 to 89.35] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 40: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group over Year 9; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 75.86, 95% CI 2-sided [43.69 to 91.07] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 41: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group over Year 10; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 71.70, 95% CI 2-sided [49.03 to 85.18] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 42: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group over Year 10; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 100.00, 95% CI 2-sided [77.89 to 100.00] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 43: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group over Year 10; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 90.00, 95% CI 2-sided [29.71 to 99.77] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 44: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group over Year 10; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 60.53, 95% CI 2-sided [26.55 to 79.83] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 45: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group over Year 10; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 48.15, 95% CI 2-sided [-2.41 to 74.87] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 46: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group over Year 11; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 82.00, 95% CI 2-sided [63.03 to 92.22] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 47: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group over Year 11; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 86.67, 95% CI 2-sided [42.67 to 98.52] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 48: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group over Year 11; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 100.00, 95% CI 2-sided [65.07 to 100.00] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 49: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group over Year 11; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 79.41, 95% CI 2-sided [52.82 to 92.30] — [estimate comment as in outcome 3, analysis 4]
Statistical Analysis 50: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group over Year 11; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 72.00, 95% CI 2-sided [33.41 to 89.77] — [estimate comment as in outcome 3, analysis 5]

5. Secondary Outcome: Number of Participants Having at Least One Post-herpetic Neuralgia (PHN) Case During the Total Duration of ZOSTER-049:EXT 006-022 Study, Overall and by Age Ranges
Description: PHN is defined by the presence of HZ-associated severe worst pain persisting or appearing more than 90 days after onset of the HZ rash. Severe worst pain is defined as HZ-associated pain rated as 3 or greater on the worst pain question on the Zoster Brief Pain Inventory (ZBPI) questionnaire. The ZBPI questionnaire uses a 0 to 10 point numeric and visual intensity scale, in which 0 represents the minimum value and 10 the maximum value on the scale. The age ranges assessed were: >=50 YOA (overall), 50-59 YOA, 60-69 YOA, >=60 YOA and >=70 YOA at time of primary vaccination in ZOSTER-006/022 studies.
Time Frame: During the total duration of ZOSTER-049:EXT 006-022 study (From Month 0 to Month 72)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- LTFU+Control >=50 YOA Group: Participants >=50 YOA (at time of primary vaccination in ZOSTER-006/022 studies) who received at least one dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study, i.e., combined group of LTFU group and Control group in the current ZOSTER-049:EXT 006-022 study.
Arm/Group | LTFU+Control >=50 YOA Group | LTFU+Control 50-59 YOA Group | LTFU+Control 60-69 YOA Group | LTFU+Control >=60 YOA Group | LTFU+Control >=70 YOA Group | Historical Control >=50 YOA Group | Historical Control 50-59 YOA Group | Historical Control 60-69 YOA Group | Historical Control >=60 YOA Group | Historical Control >=70 YOA Group
Number analyzed (Participants) | 7271 | 2046 | 1243 | 5225 | 3982 | 7271 | 2046 | 1243 | 5225 | 3982
Participants | 4 | 0 | 1 | 4 | 3 | 32 | 7 | 2 | 25 | 23
Statistical Analysis 1: Comparison: LTFU+Control >=50 YOA Group vs Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of PHN between LTFU+Control >=50 YOA Group and Historical Control>=50 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 87.50, 95% CI 2-sided [64.75 to 96.79] — VE = 1 - RR. RR = the ratio of the incidence rates of LTFU+Control >=50 YOA Group over Historical Control >=50 YOA Group. The VE of HZ/su vaccine against PHN in this study was descriptively summarized by age strata and overall
Statistical Analysis 2: Comparison: LTFU+Control 50-59 YOA Group vs Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of PHN between LTFU+Control 50-59 YOA Group and Historical Control 50-59 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 100.00, 95% CI 2-sided [46.59 to 100.00] — VE = 1 - RR. RR = the ratio of the incidence rates of LTFU+Control 50-59 YOA Group over Historical Control 50-59 YOA Group. The VE of HZ/su vaccine against PHN in this study was descriptively summarized by age strata and overall
Statistical Analysis 3: Comparison: LTFU+Control 60-69 YOA Group vs Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of PHN between LTFU+Control 60-69 YOA Group and Historical Control 60-69 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 50.00, 95% CI 2-sided [-860.45 to 99.15] — VE = 1 - RR. RR = the ratio of the incidence rates of LTFU+Control 60-69 YOA Group over Historical Control 60-69 YOA Group. The VE of HZ/su vaccine against PHN in this study was descriptively summarized by age strata and overall
Statistical Analysis 4: Comparison: LTFU+Control >=60 YOA Group vs Historical Control >=60 YOA Group; Comparison of vaccine efficacy in prevention of PHN between LTFU+Control >=60 YOA Group and Historical Control >=60 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 84.00, 95% CI 2-sided [53.66 to 95.95] — VE = 1 - RR. RR = the ratio of the incidence rates of LTFU+Control >=60 YOA Group over Historical Control >=60 YOA Group. The VE of HZ/su vaccine against PHN in this study was descriptively summarized by age strata and overall
Statistical Analysis 5: Comparison: LTFU+Control >=70 YOA Group vs Historical Control >=70 YOA Group; Comparison of vaccine efficacy in prevention of PHN between LTFU+Control >=70 YOA Group and Historical Control >=70 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 86.96, 95% CI 2-sided [56.83 to 97.49] — VE = 1 - RR. RR = the ratio of the incidence rates of LTFU+Control >=70 YOA Group over Historical Control >=70 YOA Group. The VE of HZ/su vaccine against PHN in this study was descriptively summarized by age strata and overall

6. Secondary Outcome: Number of Participants Having at Least One PHN Case From One Month Post-Dose 2 in ZOSTER-006/022 Primary Studies Until the End of ZOSTER-049:EXT 006-022 Study, Overall and by Age Ranges
Description: as for outcome 5
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Placebo/Historical Control >= 60 YOA Group: Participants between >=60 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) from the Placebo groups in the ZOSTER-006/022 primary studies for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start and from the hypothetical Historical control group in the current ZOSTER-049:EXT 006-022 study for Year 6 and onwards were combined into this group.
Arm/Group | HZ/su >=50 YOA Group | HZ/su 50-59 YOA Group | HZ/su 60-69 YOA Group | HZ/su >=60 YOA Group | HZ/su >=70 YOA Group | Placebo/Historical Control >=50 YOA Group | Placebo/Historical Control 50-59 YOA Group | Placebo/Historical Control 60-69 YOA Group | Placebo/Historical Control >= 60 YOA Group | Placebo/Historical Control >=70 YOA Group
Number analyzed (Participants) | 13881 | 3491 | 2140 | 10390 | 8250 | 14035 | 3523 | 2166 | 10512 | 8346
Participants | 8 | 0 | 1 | 8 | 7 | 78 | 15 | 4 | 63 | 59
Statistical Analysis 1: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of PHN between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 89.69, 95% CI 2-sided [78.67 to 95.70] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su >=50 YOA Group over Placebo/Historical Control >=50 YOA Group. The VE of HZ/su vaccine against PHN in this study was descriptively summarized by age strata and overall
Statistical Analysis 2: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of PHN between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 100.00, 95% CI 2-sided [77.79 to 100.00] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su 50-59 YOA Group over Placebo/Historical Control 50-59 YOA Group. The VE of HZ/su vaccine against PHN in this study was descriptively summarized by age strata and overall
Statistical Analysis 3: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of PHN between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 74.75, 95% CI 2-sided [-155.17 to 99.49] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su 60-69 YOA Group over Placebo/Historical Control 60-69 YOA Group. The VE of HZ/su vaccine against PHN in this study was descriptively summarized by age strata and overall
Statistical Analysis 4: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of PHN between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 87.24, 95% CI 2-sided [73.29 to 94.72] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su >=60 YOA Group over Placebo/Historical Control >=60 YOA Group. The VE of HZ/su vaccine against PHN in this study was descriptively summarized by age strata and overall
Statistical Analysis 5: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of PHN between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 88.08, 95% CI 2-sided [73.87 to 95.41] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su >=70 YOA Group over Placebo/Historical Control >=70 YOA Group. The VE of HZ/su vaccine against PHN in this study was descriptively summarized by age strata and overall

7. Secondary Outcome: Number of Participants Having at Least One HZ Related Complications (Other Than PHN) Case During the Total Duration of ZOSTER-049:EXT 006-022 Study, Overall and by Age Ranges
Description: HZ complications include HZ vasculitis, disseminated disease, ophthalmic disease, neurologic disease, visceral disease or stroke. If a recorded complication was associated with a case of suspected HZ, and that case was finally not considered to be a confirmed case, the associated complication would not be considered as a complication of HZ. The age ranges assessed were: >=50 YOA (overall), 50-59 YOA, 60-69 YOA, >=60 YOA and >=70 YOA at time of primary vaccination in ZOSTER-006/022 studies.
Time Frame: During the total duration of ZOSTER-049:EXT 006-022 study (From Month 0 to Month 72)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LTFU+Control >=50 YOA Group | LTFU+Control 50-59 YOA Group | LTFU+Control 60-69 YOA Group | LTFU+Control >=60 YOA Group | LTFU+Control >=70 YOA Group | Historical Control >=50 YOA Group | Historical Control 50-59 YOA Group | Historical Control 60-69 YOA Group | Historical Control >=60 YOA Group | Historical Control >=70 YOA Group
Number analyzed (Participants) | 7273 | 2046 | 1243 | 5227 | 3984 | 7273 | 2046 | 1243 | 5227 | 3984
Participants | 1 | 0 | 0 | 1 | 1 | 12 | 0 | 2 | 11 | 9
Statistical Analysis 1: Comparison: LTFU+Control >=50 YOA Group vs Historical Control >=50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ related complications between LTFU+Control >=50 YOA Group and Historical Control >=50 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 91.67, 95% CI 2-sided [43.68 to 99.81] — VE=1-RR. RR=the ratio of the incidence rates of LTFU+Control >=50 YOA Group over Historical Control >=50 YOA Group. The VE of HZ/su vaccine against HZ related complications in this study was descriptively summarized by age strata and overall
Statistical Analysis 2: Comparison: LTFU+Control 60-69 YOA Group vs Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ related complications between LTFU+Control 60-69 YOA Group and Historical Control 60-69 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 100.00, 95% CI 2-sided [-247.21 to 100.00] — VE=1-RR. RR=the ratio of the incidence rates of LTFU+Control 60-69YOA Group over Historical Control 60-69YOA Group. The VE of HZ/su vaccine against HZ related complications in this study was descriptively summarized by age strata and overall
Statistical Analysis 3: Comparison: LTFU+Control >=60 YOA Group vs Historical Control >=60 YOA Group; Comparison of vaccine efficacy in prevention of HZ related complications between LTFU+Control >=60 YOA Group and Historical Control >=60 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 90.91, 95% CI 2-sided [37.45 to 99.79] — VE=1-RR. RR=the ratio of the incidence rates of LTFU+Control >=60YOA Group over Historical Control >=60YOA Group. The VE of HZ/su vaccine against HZ related complications in this study was descriptively summarized by age strata and overall
Statistical Analysis 4: Comparison: LTFU+Control >=70 YOA Group vs Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ related complications between LTFU+Control >=70 YOA Group and Historical Control >=70 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 88.89, 95% CI 2-sided [19.81 to 99.75] — VE=1-RR. RR=the ratio of the incidence rates of LTFU+Control >=70YOA Group over Historical Control >=70YOA Group. The VE of HZ/su vaccine against HZ related complications in this study was descriptively summarized by age strata and overall

8. Secondary Outcome: Number of Participants Having at Least One HZ Related Complications (Other Than PHN) Case From One Month Post-dose 2 (Month 3) in ZOSTER-006/022 Primary Studies Until the End of ZOSTER-049:EXT 006-022 Study, Overall and by Age Ranges
Description: as for outcome 7
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- HZ/su 60-69 YOA Group: Participants between 60 to 69 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received 2 doses of the HZ/su vaccine in the ZOSTER-006/022 primary studies, among which participants who did not enroll in the current ZOSTER-049:EXT 006-022 study only contributed to data for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start.
- Placebo/Historical Control >= 50 YOA Group: Participants >=50 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) from the Placebo groups in the ZOSTER-006/022 primary studies for Year 1 through Year 4 preceding the ZOSTER-049 EXT:006-022 study start and from the hypothetical Historical control group in the current ZOSTER-049:EXT 006-022 study for Year 6 and onwards were combined into this group.
Arm/Group | HZ/su >=50 YOA Group | HZ/su 50-59 YOA Group | HZ/su 60-69 YOA Group | HZ/su >=60 YOA Group | HZ/su >=70 YOA Group | Placebo/Historical Control >= 50 YOA Group | Placebo/Historical Control 50-59 YOA Group | Placebo/Historical Control 60-69 YOA Group | Placebo/Historical Control >= 60 YOA Group | Placebo/Historical Control >=70 YOA Group
Number analyzed (Participants) | 13881 | 3491 | 2140 | 10390 | 8250 | 14035 | 3523 | 2166 | 10512 | 8346
Participants | 2 | 0 | 0 | 2 | 2 | 28 | 1 | 5 | 26 | 21
Statistical Analysis 1: Comparison: HZ/su >=50 YOA Group vs Placebo/Historical Control >= 50 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ related complications between HZ/su >=50 YOA Group and Placebo/Historical Control >=50 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 92.83, 95% CI 2-sided [71.57 to 99.17] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su >=50 YOA Group over Placebo/Historical Control >=50 YOA Group. The VE of HZ/su vaccine against HZ related complications in this study was descriptively summarized by age strata and overall
Statistical Analysis 2: Comparison: HZ/su 50-59 YOA Group vs Placebo/Historical Control 50-59 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ related complications between HZ/su 50-59 YOA Group and Placebo/Historical Control 50-59 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 100.00, 95% CI 2-sided [-1830.98 to 100.00] — VE=1-RR. RR=the ratio of the incidence rates of HZ/su 50-59YOA Group over Placebo/Historical Control 50-59YOA Group. The VE of HZ/su vaccine against HZ related complications in this study was descriptively summarized by age strata and overall
Statistical Analysis 3: Comparison: HZ/su 60-69 YOA Group vs Placebo/Historical Control 60-69 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ related complications between HZ/su 60-69 YOA Group and Placebo/Historical Control 60-69 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 100.00, 95% CI 2-sided [17.55 to 100.00] — VE=1-RR. RR=the ratio of the incidence rates of HZ/su 60-69YOA Group over Placebo/Historical Control 60-69YOA Group. The VE of HZ/su vaccine against HZ related complications in this study was descriptively summarized by age strata and overall
Statistical Analysis 4: Comparison: HZ/su >=60 YOA Group vs Placebo/Historical Control >= 60 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ related complications between HZ/su >=60 YOA Group and Placebo/Historical Control >=60 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 92.28, 95% CI 2-sided [69.17 to 99.11] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su >=60 YOA Group over Placebo/Historical Control >=60 YOA Group. The VE of HZ/su vaccine against HZ related complications in this study was descriptively summarized by age strata and overall
Statistical Analysis 5: Comparison: HZ/su >=70 YOA Group vs Placebo/Historical Control >=70 YOA Group; Comparison of vaccine efficacy (VE) in prevention of HZ related complications between HZ/su >=70 YOA Group and Placebo/Historical Control >=70 YOA Group; Test type: Other — [test comment as in outcome 1, analysis 1]; Poisson regression method; Vaccine efficacy = 90.45, 95% CI 2-sided [60.93 to 98.91] — VE = 1 - RR. RR = the ratio of the incidence rates of HZ/su >=70 YOA Group over Placebo/Historical Control >=70 YOA Group. The VE of HZ/su vaccine against HZ related complications in this study was descriptively summarized by age strata and overall

9. Secondary Outcome: Anti-glycoprotein (gE) Antibody Concentrations for Humoral Immunity (HI) Subset at Years 5, 6, 7, 8, 9, 10, 11 and 12 After the Primary Vaccination in ZOSTER-006/022 Studies, Overall and by Age Ranges in the LTFU Group
Description: Anti-gE antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs) in milli-international units per milliliter (mIU/mL). The age ranges assessed were: >=50 YOA (overall), 50-59 YOA, 60-69 YOA, >=60 YOA and >=70 YOA at time of primary vaccination in ZOSTER-006/022 studies.
Time Frame: At Years 5, 6, 7, 8, 9, 10, 11 and 12 after the primary vaccination in ZOSTER-006/022 studies
Population: The analysis was performed on a subset of participants from the Adapted ATP cohort for humoral persistence - LTFU, who were included in the immunogenicity subset during the ZOSTER-006/022 studies, continued participation in this study and had humoral persistence results available at the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Groups:
- LTFU >=50 YOA Group: Participants >=50 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received at least 1 dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study.
- LTFU 50-59 YOA Group: Participants between 50 and 59 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received at least 1 dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study.
- LTFU 60-69 YOA Group: Participants between 60 and 69 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received at least 1 dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study.
- LTFU >=60 YOA Group: Participants >=60 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received at least 1 dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study.
- LTFU >=70 YOA Group: Participants >=70 YOA (at the time of primary vaccination in ZOSTER-006/022 studies) who received at least 1 dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study.
Arm/Group | LTFU >=50 YOA Group | LTFU 50-59 YOA Group | LTFU 60-69 YOA Group | LTFU >=60 YOA Group | LTFU >=70 YOA Group
Number analyzed (Participants) | 786 | 219 | 230 | 567 | 337
mIU/mL
  Year 5: number analyzed (Participants) | 214 | 51 | 35 | 163 | 128
  Year 5 | 8043.5 [7224.9 to 8954.7] | 8044.2 [6106.6 to 10596.6] | 8715.1 [6807.0 to 11158.1] | 8043.2 [7180.7 to 9009.3] | 7868.7 [6915.4 to 8953.5]
  Year 6 | 8536.6 [8113.5 to 8981.7] | 8584.3 [7739.9 to 9520.7] | 8913.4 [8155.1 to 9742.3] | 8518.3 [8036.5 to 9028.9] | 8258.7 [7646.0 to 8920.4]
  Year 7: number analyzed (Participants) | 757 | 215 | 222 | 542 | 320
  Year 7 | 8375.1 [7941.0 to 8833.0] | 8325.6 [7483.0 to 9263.1] | 8869.6 [8084.4 to 9731.1] | 8394.8 [7895.3 to 8925.8] | 8080.4 [7446.1 to 8768.7]
  Year 8: number analyzed (Participants) | 732 | 215 | 219 | 517 | 298
  Year 8 | 8231.2 [7778.2 to 8710.6] | 8318.0 [7412.7 to 9333.9] | 8680.0 [7901.2 to 9535.5] | 8195.4 [7683.4 to 8741.5] | 7856.6 [7193.3 to 8581.0]
  Year 9: number analyzed (Participants) | 641 | 199 | 195 | 442 | 247
  Year 9 | 7219.4 [6803.4 to 7660.9] | 7097.6 [6341.6 to 7943.7] | 7706.7 [6994.6 to 8491.4] | 7275.0 [6784.2 to 7801.3] | 6951.3 [6295.8 to 7674.9]
  Year 10: number analyzed (Participants) | 606 | 197 | 187 | 409 | 222
  Year 10 | 6861.5 [6433.2 to 7318.3] | 7007.0 [6228.4 to 7882.9] | 7060.8 [6304.2 to 7908.3] | 6792.5 [6288.2 to 7337.3] | 6574.4 [5913.8 to 7308.8]
  Year 11: number analyzed (Participants) | 612 | 196 | 192 | 416 | 224
  Year 11 | 7039.3 [6589.0 to 7520.5] | 7146.9 [6294.9 to 8114.3] | 7159.8 [6406.3 to 8001.9] | 6989.2 [6470.8 to 7549.2] | 6846.3 [6148.5 to 7623.3]
  Year 12: number analyzed (Participants) | 435 | 151 | 161 | 284 | 123
  Year 12 | 6844.3 [6335.2 to 7394.3] | 6737.1 [5900.9 to 7691.7] | 6943.4 [6071.3 to 7940.7] | 6902.0 [6272.0 to 7595.3] | 6848.2 [5976.0 to 7847.6]

10. Secondary Outcome: Frequency of Antigen-specific CD4 (2+) T-cells for Cell Mediated Immunity (CMI) Subset at Years 5, 6, 7, 8, 9, 10, 11 and 12 After the Primary Vaccination in ZOSTER-006/022 Studies, Overall and by Age Ranges in the LTFU Group
Description: Frequency of CD4 (2+) T-cells with antigen-specific Interferon gamma (IFN-γ) and/or Interleukin-2 (IL-2) and/or Tumour Necrosis Factor alpha (TNF-α) and/or CD40 Ligand (CD40L) secretion/expression to gE was determined by Intracellular Cytokine Staining (ICS) and expressed in CD4 (2+) T-cells/million cells. The age ranges assessed were: >=50 YOA (overall), 50-59 YOA, 60-69 YOA, >=60 YOA and >=70 YOA at time of primary vaccination in ZOSTER-006/022 studies.
Time Frame: At Years 5, 6, 7, 8, 9, 10, 11 and 12 after the primary vaccination in ZOSTER-006/022 studies
Population: The analysis was performed on a subset of participants from the Adapted ATP cohort for CMI persistence - LTFU, who were included in the CMI subset during ZOSTER-006/-022 studies, continued participation in this study and had CMI results available at the specified time points.
Measure: Mean (Standard Deviation); unit: CD4 (2+) T-cells/million cells
Arm/Group | LTFU >=50 YOA Group | LTFU 50-59 YOA Group | LTFU 60-69 YOA Group | LTFU >=60 YOA Group | LTFU >=70 YOA Group
Number analyzed (Participants) | 100 | 39 | 38 | 61 | 24
CD4 (2+) T-cells/million cells
  Year 5: number analyzed (Participants) | 3 | 2 | 0 | 1 | 1
  Year 5 | 698.00 (531.11) | 858.92 (639.37) |  | 376.16 (NA) — Standard deviation could not be calculated as there was only one participant with frequency of antigen-specific CD4 (2+) T-cells data available. | 376.16 (NA) — Standard deviation could not be calculated as there was only one participant with frequency of antigen-specific CD4 (2+) T-cells data available.
  Year 6: number analyzed (Participants) | 100 | 39 | 38 | 61 | 23
  Year 6 | 886.15 (869.09) | 1174.70 (1103.76) | 839.31 (644.97) | 701.66 (621.26) | 474.23 (515.96)
  Year 7: number analyzed (Participants) | 100 | 39 | 37 | 61 | 24
  Year 7 | 859.46 (881.80) | 1141.00 (1074.96) | 745.36 (572.57) | 679.46 (683.15) | 577.87 (828.60)
  Year 8: number analyzed (Participants) | 97 | 37 | 38 | 60 | 22
  Year 8 | 896.26 (925.58) | 1217.84 (1155.53) | 737.78 (602.91) | 697.96 (688.76) | 629.18 (827.35)
  Year 9: number analyzed (Participants) | 84 | 34 | 35 | 50 | 15
  Year 9 | 1099.20 (1151.15) | 1403.78 (1435.49) | 930.89 (796.20) | 892.09 (865.29) | 801.54 (1033.67)
  Year 10: number analyzed (Participants) | 80 | 35 | 31 | 45 | 14
  Year 10 | 1016.13 (992.38) | 1210.28 (1216.92) | 952.86 (763.05) | 865.13 (755.35) | 670.87 (726.96)
  Year 11: number analyzed (Participants) | 83 | 36 | 33 | 47 | 14
  Year 11 | 909.95 (1025.40) | 1113.90 (1317.91) | 884.65 (712.45) | 753.74 (703.75) | 445.15 (597.48)
  Year 12: number analyzed (Participants) | 73 | 32 | 29 | 41 | 12
  Year 12 | 853.77 (815.20) | 1030.37 (971.86) | 828.62 (666.18) | 715.95 (647.90) | 443.65 (531.44)

11. Secondary Outcome: Anti-gE Antibody Concentrations for Participants in LTFU+Control >=50 YOA Group (With a Confirmed HZ Episode) at Years 5, 6, 7, 8, 9, 10, 11 and 12 After the Primary Vaccination in ZOSTER-006/022 Studies
Description: Anti-gE antibody concentrations were determined by ELISA and expressed as GMCs in mIU/mL.
Time Frame: At Years 5, 6, 7, 8, 9, 10, 11 and 12 after the primary vaccination in ZOSTER-006/022 studies
Population: The analysis was performed on a HZ subset for HI, which included participants who developed confirmed HZ during ZOSTER-006 or ZOSTER-022 studies, or who developed HZ during the interval between the end of the ZOSTER-006/022 studies and the beginning of the current ZOSTER-049:EXT 006-022 study, or who developed suspected HZ during the current ZOSTER-049:EXT 006-022 study and with immunogenicity results available for the specified analysis at the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Groups:
- LTFU+Control >=50 YOA Group: Participants >=50 YOA (at the time of primary vaccination in the ZOSTER-006/022 studies) who received at least one dose of the HZ/su vaccine in the ZOSTER-006/022 primary studies and no additional doses of the HZ/su vaccine in the current ZOSTER-049:EXT 006-022 study, i.e., combined group of LTFU group and Control group in the current ZOSTER-049:EXT 006-022 study.
Arm/Group | LTFU+Control >=50 YOA Group
Number analyzed (Participants) | 62
mIU/mL
  Year 5: number analyzed (Participants) | 6
  Year 5 | 12455.1 [8549.9 to 18144.1]
  Year 6: number analyzed (Participants) | 22
  Year 6 | 8138.7 [5770.6 to 11478.7]
  Year 7: number analyzed (Participants) | 30
  Year 7 | 6888.0 [4919.2 to 9644.7]
  Year 8: number analyzed (Participants) | 39
  Year 8 | 5831.9 [4435.1 to 7668.6]
  Year 9: number analyzed (Participants) | 38
  Year 9 | 7706.8 [5941.6 to 9996.5]
  Year 10: number analyzed (Participants) | 48
  Year 10 | 6800.1 [5048.6 to 9159.2]
  Year 11 | 6214.7 [4807.3 to 8034.2]
  Year 12: number analyzed (Participants) | 30
  Year 12 | 4770.7 [3523.6 to 6459.2]

12. Secondary Outcome: Frequency of Antigen-specific CD4 (2+) T-cells for Participants in LTFU+Control >=50 YOA Group (With a Confirmed HZ Episode) at Years 5, 6, 7, 8, 9 and 10 After the Primary Vaccination in ZOSTER-006/022 Studies
Description: Frequency of CD4 (2+) T-cells with antigen-specific IFN-γ and/or IL-2 and/or TNF-α and/or CD40L secretion/expression to gE was determined by ICS and expressed in CD4 (2+) T-cells/million cells.
Time Frame: At Years 5, 6, 7, 8, 9, and 10 after the primary vaccination in ZOSTER-006/022 studies
Population: The analysis was performed on a HZ subset for CMI, which included participants who developed confirmed HZ during ZOSTER-006 or ZOSTER-022 studies, or who developed HZ during the interval between the end of the ZOSTER-006/022 studies and the beginning of the current ZOSTER-049:EXT 006-022 study, or who developed suspected HZ during the current ZOSTER-049:EXT 006-022 study and with CMI results available for the specified analysis at the specified time points.
Measure: Mean (Standard Deviation); unit: CD4 (2+) T-cells/million cells
Arm/Group | LTFU+Control >=50 YOA Group
Number analyzed (Participants) | 2
CD4 (2+) T-cells/million cells
  Year 5: number analyzed (Participants) | 1
  Year 5 | 683.76 (NA) — Standard deviation could not be calculated as there was only one participant with frequency of antigen-specific CD4 (2+) T-cells data available.
  Year 6 | 398.70 (164.34)
  Year 7 | 347.43 (138.41)
  Year 8: number analyzed (Participants) | 1
  Year 8 | 509.67 (NA) — Standard deviation could not be calculated as there was only one participant with frequency of antigen-specific CD4 (2+) T-cells data available.
  Year 10: number analyzed (Participants) | 1
  Year 10 | 749.75 (NA) — Standard deviation could not be calculated as there was only one participant with frequency of antigen-specific CD4 (2+) T-cells data available.

13. Secondary Outcome: Anti-gE Antibody Concentrations for 1-Additional Dose, Revaccination and Control Groups at Month 1 in the Current ZOSTER-049:EXT 006-022 Study
Description: Anti-gE antibody concentrations were determined by ELISA and expressed as GMCs in mIU/mL.
Time Frame: At Month 1 in the current ZOSTER-049:EXT 006-022 study
Population: Adapted ATP cohort for immunogenicity included all participants who met all eligibility criteria, received all doses as per assignment*, for whom administration site of study vaccine was known*, who did not receive any other vaccine, who complied with the procedures defined in protocol, vaccination* and blood sample schedule and with immunogenicity data available for the specified analysis at the specified time point.
  *only applicable for the participants revaccinated in the current study.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 1-Additional Dose Group | Revaccination Group | Control Group
Number analyzed (Participants) | 58 | 55 | 117
mIU/mL | 73834.4 [60603.6 to 89953.7] | 79419.8 [65089.6 to 96904.9] | 9655.2 [8316.9 to 11208.8]

14. Secondary Outcome: Frequency of Antigen-specific CD4(2+) T-cells for 1-Additional Dose, Revaccination and Control Groups at Month 1 in the Current ZOSTER-049:EXT 006-022 Study
Description: as for outcome 12
Time Frame: At Month 1 in the current ZOSTER-049:EXT 006-022 study
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: CD4 (2+) T-cells/million cells
Arm/Group | 1-Additional Dose Group | Revaccination Group | Control Group
Number analyzed (Participants) | 52 | 46 | 104
CD4 (2+) T-cells/million cells | 3899.69 (3243.16) | 2803.96 (1544.14) | 716.01 (635.32)

15. Secondary Outcome: Anti-gE Antibody Concentrations for Revaccination and Control Groups at Month 3 in the Current ZOSTER-049:EXT 006-022 Study
Description: Anti-gE antibody concentrations were determined by ELISA and expressed as GMCs in mIU/mL.
Time Frame: At Month 3 in the current ZOSTER-049:EXT 006-022 study
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Revaccination Group | Control Group
Number analyzed (Participants) | 55 | 117
mIU/mL | 64603.0 [54008.4 to 77275.9] | 9428.1 [8154.4 to 10900.8]

16. Secondary Outcome: Frequency of Antigen-specific CD4 (2+) T-cells for Revaccination and Control Groups at Month 3 in the Current ZOSTER-049:EXT 006-022 Study
Description: as for outcome 12
Time Frame: At Month 3 in the current ZOSTER-049:EXT 006-022 study
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: CD4 (2+) T-cells/million cells
Arm/Group | Revaccination Group | Control Group
Number analyzed (Participants) | 51 | 107
CD4 (2+) T-cells/million cells | 2443.17 (3896.14) | 739.07 (659.78)

17. Secondary Outcome: Anti-gE Antibody Concentrations for 1 Additional Dose, Revaccination and Control Groups at Month 0 and Years 1, 2, 3, 4, 5 and 6 in the Current ZOSTER-049:EXT 006-022 Study
Description: Anti-gE antibody concentrations were determined by ELISA and expressed as GMCs in mIU/mL.
Time Frame: At Month 0 and Years 1, 2, 3, 4, 5 and 6 in the current ZOSTER-049:EXT 006-022 study
Population: Adapted ATP cohort for immunogenicity included all participants who met all eligibility criteria, received all doses as per assignment*, for whom administration site of study vaccine was known*, who did not receive any other vaccine, who complied with the procedures defined in protocol, vaccination* and blood sample schedule and with immunogenicity data available for the specified analysis at the specified time points.
  *only applicable for the participants revaccinated in the current study.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 1-Additional Dose Group | Revaccination Group | Control Group
Number analyzed (Participants) | 60 | 55 | 117
mIU/mL
  Month 0: number analyzed (Participants) | 58 | 55 | 117
  Month 0 | 10149.5 [8640.2 to 11922.4] | 11548.5 [9386.8 to 14208.0] | 10232.0 [8836.7 to 11847.5]
  Year 1: number analyzed (Participants) | 60 | 52 | 115
  Year 1 | 24663.6 [20790.2 to 29258.7] | 26167.5 [21755.6 to 31474.2] | 8825.4 [7616.3 to 10226.5]
  Year 2: number analyzed (Participants) | 59 | 51 | 112
  Year 2 | 19417.9 [16460.7 to 22906.4] | 19973.2 [16538.1 to 24121.8] | 8643.3 [7450.5 to 10027.0]
  Year 3: number analyzed (Participants) | 57 | 51 | 108
  Year 3 | 16335.6 [13890.4 to 19211.3] | 16264.7 [13417.7 to 19715.7] | 8314.9 [7080.3 to 9764.7]
  Year 4: number analyzed (Participants) | 48 | 44 | 94
  Year 4 | 18676.4 [15562.0 to 22414.2] | 16363.2 [13219.3 to 20254.9] | 8581.7 [7195.2 to 10235.3]
  Year 5: number analyzed (Participants) | 52 | 47 | 99
  Year 5 | 14797.3 [12340.7 to 17742.9] | 14595.7 [11767.0 to 18104.4] | 7238.7 [6004.3 to 8727.0]
  Year 6: number analyzed (Participants) | 50 | 46 | 91
  Year 6 | 12868.4 [11048.3 to 14988.2] | 13534.0 [11107.7 to 16490.2] | 6858.8 [5698.0 to 8256.3]

18. Secondary Outcome: Frequency of Antigen-specific CD4(2+) T-cells for 1-Additional Dose, Revaccination and Control Groups at Month 0 and Years 1, 2, 3, 4, 5 and 6 in the Current ZOSTER-049:EXT 006-022 Study
Description: as for outcome 12
Time Frame: At Month 0 and Years 1, 2, 3, 4, 5 and 6 in the current ZOSTER-049:EXT 006-022 study
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: CD4(2+) T-cells/million cells
Arm/Group | 1-Additional Dose Group | Revaccination Group | Control Group
Number analyzed (Participants) | 58 | 54 | 109
CD4(2+) T-cells/million cells
  Month 0: number analyzed (Participants) | 55 | 54 | 109
  Month 0 | 843.55 (792.93) | 876.23 (784.84) | 817.97 (809.77)
  Year 1: number analyzed (Participants) | 53 | 50 | 97
  Year 1 | 1798.39 (2119.46) | 1155.04 (714.97) | 665.50 (603.93)
  Year 2: number analyzed (Participants) | 58 | 46 | 109
  Year 2 | 1634.47 (1900.93) | 1154.97 (818.16) | 712.02 (715.32)
  Year 3: number analyzed (Participants) | 51 | 45 | 95
  Year 3 | 2112.90 (2564.29) | 1219.13 (889.76) | 836.62 (921.57)
  Year 4: number analyzed (Participants) | 45 | 43 | 83
  Year 4 | 2047.92 (2477.92) | 1083.64 (669.54) | 901.57 (917.41)
  Year 5: number analyzed (Participants) | 48 | 47 | 93
  Year 5 | 1649.03 (2407.72) | 917.93 (648.92) | 720.32 (726.20)
  Year 6: number analyzed (Participants) | 48 | 41 | 82
  Year 6 | 1682.94 (2694.90) | 844.81 (651.28) | 736.01 (724.10)

19. Secondary Outcome: Number of Participants With Any and Grade 3 Solicited Local Symptoms
Description: The assessed solicited local symptoms included pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within 7 days after each vaccination (vaccination occurring at Month 0 for 1-Additional Dose Group and at Months 0 and 2 for Revaccination Group) in the current ZOSTER-049:EXT 006-022 study
Population: The analysis was performed on the Total Vaccinated Cohort (for 1-Additional Dose and Revaccination groups), which included all participants who received at least 1 dose of the study treatment in ZOSTER-049:EXT 006-022 study and who have documented solicited symptoms (i.e., diary card for solicited AEs completed and returned) after each vaccination. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Additional Dose Group | Revaccination Group
Number analyzed (Participants) | 61 | 60
Participants
  Any pain, post-Dose 1 | 42 | 52
  Grade 3 pain, post-Dose 1 | 1 | 3
  Any redness, post-Dose 1 | 13 | 20
  Grade 3 redness, post-Dose 1 | 4 | 1
  Any swelling, post-Dose 1 | 7 | 12
  Grade 3 swelling, post-Dose 1 | 1 | 0
  Any pain, post-Dose 2: number analyzed (Participants) | 0 | 55
  Any pain, post-Dose 2 |  | 37
  Grade 3 pain, post-Dose 2: number analyzed (Participants) | 0 | 55
  Grade 3 pain, post-Dose 2 |  | 2
  Any redness, post-Dose 2: number analyzed (Participants) | 0 | 55
  Any redness, post-Dose 2 |  | 20
  Grade 3 redness, post-Dose 2: number analyzed (Participants) | 0 | 55
  Grade 3 redness, post-Dose 2 |  | 3
  Any swelling, post-Dose 2: number analyzed (Participants) | 0 | 55
  Any swelling, post-Dose 2 |  | 13
  Grade 3 swelling, post-Dose 2: number analyzed (Participants) | 0 | 55
  Grade 3 swelling, post-Dose 2 |  | 1

20. Secondary Outcome: Duration in Days of Solicited Local Symptoms
Description: Duration is the number of days in which a participant experienced the symptom within the 7-day solicited follow-up period. The assessed solicited local symptoms included pain, redness and swelling.
Time Frame: as for outcome 19
Population: The analysis was performed on the Total Vaccinated Cohort (for 1-Additional Dose and Revaccination groups), which included all participants who received at least 1 dose of the study treatment in ZOSTER-049:EXT 006-022 study, with diary data available after each vaccination and who experienced the specified solicited local symptom within 7 days following the respective vaccine dose. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 1-Additional Dose Group | Revaccination Group
Number analyzed (Participants) | 61 | 60
Days
  Pain, post-Dose 1 | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 3.5]
  Pain, post-Dose 2: number analyzed (Participants) | 0 | 55
  Pain, post-Dose 2 |  | 2.0 [2.0 to 3.0]
  Redness, post-Dose 1 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Redness, post-Dose 2: number analyzed (Participants) | 0 | 55
  Redness, post-Dose 2 |  | 2.5 [1.0 to 4.5]
  Swelling, post-Dose 1 | 2.0 [2.0 to 3.0] | 3.0 [1.0 to 5.0]
  Swelling, post-Dose 2: number analyzed (Participants) | 0 | 55
  Swelling, post-Dose 2 |  | 2.0 [1.0 to 3.0]

21. Secondary Outcome: Number of Participants With Any, Grade 3 and Related Solicited General Symptoms
Description: The assessed solicited general symptoms included fatigue, fever [defined as oral temperature >=37.5 degrees Celsius (°C)], gastrointestinal symptoms, headache, myalgia, and shivering. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever >39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Additional Dose Group | Revaccination Group
Number analyzed (Participants) | 61 | 60
Participants
  Any fatigue, post-Dose 1 | 32 | 24
  Grade 3 fatigue, post-Dose 1 | 0 | 2
  Related fatigue, post-Dose 1 | 32 | 23
  Any fever, post-Dose 1 | 18 | 13
  Grade 3 fever, post-Dose 1 | 0 | 0
  Related fever, post-Dose 1 | 18 | 13
  Any gastrointestinal symptoms, post-Dose 1 | 9 | 9
  Grade 3 gastrointestinal symptoms, post-Dose 1 | 0 | 2
  Related gastrointestinal symptoms, post-Dose 1 | 9 | 8
  Any headache, post-Dose 1 | 23 | 17
  Grade 3 headache, post-Dose 1 | 0 | 2
  Related headache, post-Dose 1 | 23 | 17
  Any myalgia, post-Dose 1 | 27 | 22
  Grade 3 myalgia, post-Dose 1 | 0 | 2
  Related myalgia, post-Dose 1 | 27 | 21
  Any shivering, post-Dose 1 | 25 | 15
  Grade 3 shivering, post-Dose 1 | 2 | 4
  Related shivering, post-Dose 1 | 25 | 15
  Any fatigue, post-Dose 2: number analyzed (Participants) | 0 | 55
  Any fatigue, post-Dose 2 |  | 22
  Grade 3 fatigue, post-Dose 2: number analyzed (Participants) | 0 | 55
  Grade 3 fatigue, post-Dose 2 |  | 3
  Related fatigue, post-Dose 2: number analyzed (Participants) | 0 | 55
  Related fatigue, post-Dose 2 |  | 21
  Any fever, post-Dose 2: number analyzed (Participants) | 0 | 55
  Any fever, post-Dose 2 |  | 7
  Grade 3 fever, post-Dose 2: number analyzed (Participants) | 0 | 55
  Grade 3 fever, post-Dose 2 |  | 0
  Related fever, post-Dose 2: number analyzed (Participants) | 0 | 55
  Related fever, post-Dose 2 |  | 4
  Any gastrointestinal symptoms, post-Dose 2: number analyzed (Participants) | 0 | 55
  Any gastrointestinal symptoms, post-Dose 2 |  | 4
  Grade 3 gastrointestinal symptoms, post-Dose 2: number analyzed (Participants) | 0 | 55
  Grade 3 gastrointestinal symptoms, post-Dose 2 |  | 0
  Related gastrointestinal symptoms, post-dose 2: number analyzed (Participants) | 0 | 55
  Related gastrointestinal symptoms, post-dose 2 |  | 4
  Any headache, post-Dose 2: number analyzed (Participants) | 0 | 55
  Any headache, post-Dose 2 |  | 15
  Grade 3 headache, post-Dose 2: number analyzed (Participants) | 0 | 55
  Grade 3 headache, post-Dose 2 |  | 1
  Related headache, post-Dose 2: number analyzed (Participants) | 0 | 55
  Related headache, post-Dose 2 |  | 14
  Any myalgia, post-Dose 2: number analyzed (Participants) | 0 | 55
  Any myalgia, post-Dose 2 |  | 12
  Grade 3 myalgia, post-Dose 2: number analyzed (Participants) | 0 | 55
  Grade 3 myalgia, post-Dose 2 |  | 1
  Related myalgia, post-Dose 2: number analyzed (Participants) | 0 | 55
  Related myalgia, post-Dose 2 |  | 11
  Any shivering, post-Dose 2: number analyzed (Participants) | 0 | 55
  Any shivering, post-Dose 2 |  | 7
  Grade 3 shivering, post-Dose 2: number analyzed (Participants) | 0 | 55
  Grade 3 shivering, post-Dose 2 |  | 0
  Related shivering, post-Dose 2: number analyzed (Participants) | 0 | 55
  Related shivering, post-Dose 2 |  | 7

22. Secondary Outcome: Duration in Days of Solicited General Symptoms
Description: Duration is the number of days in which a participant experienced the symptom within the 7-day solicited follow-up period. The assessed solicited general symptoms included fatigue, fever [defined as oral temperature >=37.5°C], gastrointestinal symptoms, headache, myalgia, and shivering.
Time Frame: as for outcome 19
Population: The analysis was performed on the Total Vaccinated Cohort (for 1-Additional Dose and Revaccination groups), which included all participants who received at least 1 dose of the study treatment in ZOSTER-049:EXT 006-022 study, with diary data available after each vaccination and who experienced the specified solicited general symptom within 7 days following the respective vaccine dose. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 1-Additional Dose Group | Revaccination Group
Number analyzed (Participants) | 61 | 60
Days
  Fatigue, post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Fatigue, post-Dose 2: number analyzed (Participants) | 0 | 55
  Fatigue, post-Dose 2 |  | 2.0 [1.0 to 3.0]
  Fever, post-Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Fever, post-Dose 2: number analyzed (Participants) | 0 | 55
  Fever, post-Dose 2 |  | 1.0 [1.0 to 2.0]
  Gastrointestinal symptoms, post-Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Gastrointestinal symptoms, post-Dose 2: number analyzed (Participants) | 0 | 55
  Gastrointestinal symptoms, post-Dose 2 |  | 1.5 [1.0 to 2.0]
  Headache, post-Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Headache, post-Dose 2: number analyzed (Participants) | 0 | 55
  Headache, post-Dose 2 |  | 2.0 [1.0 to 3.0]
  Myalgia, post-Dose 1 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Myalgia, post-Dose 2: number analyzed (Participants) | 0 | 55
  Myalgia, post-Dose 2 |  | 1.5 [1.0 to 2.5]
  Shivering, post-Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Shivering, post-Dose 2: number analyzed (Participants) | 0 | 55
  Shivering, post-Dose 2 |  | 1.0 [1.0 to 2.0]

23. Secondary Outcome: Number of Participants With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is defined as any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 30 days after any vaccination (vaccination occurring at Month 0 for 1-Additional Dose Group and at Months 0 and 2 for Revaccination Group) in the current ZOSTER-049:EXT 006-022 study
Population: The analysis was performed on the Total Vaccinated Cohort (for 1-Additional Dose and Revaccination groups), which included all participants who received at least 1 dose of the study treatment in ZOSTER-049:EXT 006-022 study.
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Additional Dose Group | Revaccination Group
Number analyzed (Participants) | 61 | 60
Participants | 13 | 15

24. Secondary Outcome: Number of Participants With Any and Related Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant. Any SAE = occurrence of the SAE regardless of intensity or relation to study vaccination. Related SAE = SAE assessed by the investigator as related to vaccination.
Time Frame: From Month 0 to Month 12 (1-Additional Dose and Control groups) and from Month 0 until 12 months after last HZ/su vaccination (Revaccination group)
Population: The analysis was performed on Total Vaccinated cohort, which included all participants who received at least 1 dose of the study treatment in ZOSTER-049:EXT 006-022 study (1-Additional Dose and Revaccination groups) and all participants who came for Month 0 visit (Control group).
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Additional Dose Group | Revaccination Group | Control Group
Number analyzed (Participants) | 61 | 60 | 119
Participants
  Any SAEs | 4 | 4 | 11
  Related SAEs | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With SAEs Related to Investigational Vaccine, Related to Study Participation or to GSK Concomitant Medication/Vaccine
Description: An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant.
Time Frame: During the total duration of ZOSTER-049:EXT 006-022 study (from Month 0 to Month 72)
Population: The analysis was performed on Total Vaccinated cohort, which included all participants who received at least 1 dose of the study treatment in ZOSTER-049:EXT 006-022 study (1-Additional Dose and Revaccination groups) and all participants who came for Month 0 visit (LTFU and Control groups).
Measure: Count of Participants; unit: Participants
Arm/Group | LTFU Group | 1-Additional Dose Group | Revaccination Group | Control Group
Number analyzed (Participants) | 7289 | 61 | 60 | 119
Participants | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With Any and Related Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are defined as a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Any pIMDs = occurrence of a pIMD regardless of relation to vaccination. Related pIMD = a pIMD assessed by the investigator as related to the study vaccination.
Time Frame: From Month 0 to Month 12 (1-Additional Dose and Control groups) and from Month until 12 months after last HZ/su vaccination (Revaccination group)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Additional Dose Group | Revaccination Group | Control Group
Number analyzed (Participants) | 61 | 60 | 119
Participants
  Any pIMDs | 0 | 0 | 0
  Related pIMDs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs: Within 7 days after any vaccination & Unsolicited AEs: Within 30 days after any vaccination in this study. All-cause mortality & SAEs related to investigational vaccine/study participation/GSK concomitant medication/vaccine: during the entire study period (Month 0 to Month 72) (all study groups). All SAEs: Month 0 to Month 12 (1-Additional Dose & Control groups) and Month 0 until 12 months after last HZ/su vaccination (Revaccination group).
Description: As pre-specified in protocol, data in the Other (Non-Serious) Adverse Events module was only collected for the revaccinated participants in ZOSTER-049:EXT 006-022 study (1-Additional Dose and Revaccination groups).
  As per the change in AE reporting requirements from protocol amendment 2 onwards, only the related SAEs were recorded in the electronic case report form (eCRF) for LTFU group and reported.
Arm/Group | LTFU Group | 1-Additional Dose Group | Revaccination Group | Control Group
All-Cause Mortality (participants affected / at risk) | 56/7289 | 0/61 | 0/60 | 0/119
Serious Adverse Events (participants affected / at risk) | 62/7289 | 4/61 | 4/60 | 11/119
Other Adverse Events (participants affected / at risk) | 0/0 | 54/61 | 58/60 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LTFU Group (N=7289) | 1-Additional Dose Group (N=61) | Revaccination Group (N=60) | Control Group (N=119)
Cardiac arrest (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cardiac disoder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 14 (14) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Cardiac hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adams-stokes syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LTFU Group (N=0) | 1-Additional Dose Group (N=61) | Revaccination Group (N=60) | Control Group (N=0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 9 (9) | 10 (13) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 26 (26) | 19 (22) | 0 (0)
Fatigue (General disorders) | 0 (0) | 32 (32) | 33 (46) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 42 (42) | 53 (89) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 18 (18) | 17 (20) | 0 (0)
Swelling (General disorders) | 0 (0) | 7 (7) | 16 (25) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 27 (27) | 26 (34) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 24 (25) | 23 (33) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 13 (13) | 28 (42) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT02723773/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT02723773/SAP_001.pdf